CLINICAL TRIAL: NCT01386359
Title: Evaluating Nulojix Long-Term Safety in Transplant
Brief Title: Evaluating Nulojix (Belatacept) Long-Term Safety in Transplant
Acronym: ENLIST
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-076
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult de novo EBV-seropositive kidney-transplant recipients: Adult de novo EBV-seropositive kidney-transplant recipients treated with Nulojix (belatacept)
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — No Intervention. Subjects are previously treated with Nulojix (belatacept)

SUMMARY:
To describe how Nulojix (belatacept) is used and to determine how often Post-Transplant Lymphoproliferative Disorder (PTLD), Central Nervous System (CNS) PTLD and Progressive Multifocal Leukoencephalopathy (PML), rare and serious complications of transplant treatment, occur in patients taking Nulojix (belatacept) in a real-world setting.

DETAILED DESCRIPTION:
Time Perspective: Prospective for the majority of patients who are enrolled at the time they begin Nulojix (belatacept) treatment. Retrospective for any patients receiving Nulojix (belatacept) prior to enrollment into ENLiST Registry

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant recipient (age ≥18 years at time of transplant)
* Kidney-only transplant recipient
* Positive EBV serostatus

  a) EBV serostatus negative or unknown included per the investigator discretion
* Received first dose of Nulojix (Belatacept) within ≤ 14 days of renal transplant
* Received first dose of Nulojix (Belatacept) as part of normal clinical care (i.e. not as part of a clinical trial)

Exclusion Criteria:

* Received Nulojix (belatacept) for non kidney transplants
* <18 years of age at time of transplant
* Received first dose of Nulojix (belatacept) as an assigned study drug under a clinical trial protocol
* EBV-serostatus negative or unknown patients, except by investigator decision
* Patient who did not receive Belatacept for de novo treatment
* Recipient of concurrent or extant non-kidney organ transplant
* Received first dose of Nulojix (belatacept) > 14 days after date of renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult de novo EBV-seropositive kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2012-02-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of confirmed PTLD in US adult de novo Epstein Barr Virus (EBV)-seropositive kidney transplant recipients treated with Nulojix (belatacept) in clinical practice | Every 6 months for up to 72 months
Incidence rate of confirmed CNS PTLD in US adult de novo Epstein Barr Virus (EBV)-seropositive kidney transplant recipients treated with Nulojix (belatacept) in clinical practice | Every 6 months for up to 72 months
Incidence rate of PML in confirmed PML in US adult de novo Epstein Barr Virus (EBV)-seropositive kidney transplant recipients treated with Nulojix (belatacept) in clinical practice | Every 6 months for up to 72 months

SECONDARY OUTCOMES:
Demographic, clinical and treatment characteristics of patients receiving Nulojix (belatacept) | Every 6 months for up to 72 months
Rates of graft survival observed in the Nulojix (belatacept) treated patients | Every 6 months for up to 72 months
Rates of patient survival observed in the Nulojix (belatacept) treated patients | Every 6 months for up to 72 months
Incidence rate of confirmed PTLD and confirmed CNS PTLD by baseline CMV serostatus among Nulojix (belatacept) treated population | Every 6 months for up to 72 months
Incidence rates of total reported PTLD, reported CNS PTLD and reported PML in adult de novo EBV seropositive kidney transplant recipients treated with Nulojix (belatacept) | Every 6 months for up to 72 months
Incidence rates of total reported PTLD and of total reported CNS PTLD by baseline CMV serostatus among Nulojix (belatacept) treated patients | Every 6 months for up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (36):
  - University of Arizona, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Med Center, Los Angeles, California
  - St. Vincent Medical Center - Los Angeles, Los Angeles, California
  - California Institute of Renal Research, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Denver Nephrologists, Denver, Colorado
  - Yale University (Yale New Haven Hospital), New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Emory Healthcare - Emory University Hospital (EUH), Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois Mecial Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Lutheran Kidney Transplant Center, Fort Wayne, Indiana
  - The Iowa Clinic, Des Moines, Iowa
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Clair Nephrology Research, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Bms Clinical Research Center, Does Not Exist, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York- Presbyterian/ Weill Cornell Medical Canter, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Christ Hospital Cancer Research, Cincinnati, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Univ of Virginia HSC, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm